CLINICAL TRIAL: NCT02146599
Title: Patient Perception of Visual Quality and Function
Status: Completed | Type: Observational
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Other Study IDs: QPRO-101-SIVQ
Record Dates: First submitted 2014-05-20; First posted 2014-05-26 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pseudophakic
  Interventions: Other: Administration of patient self-assessment

INTERVENTIONS:
Other: Administration of patient self-assessment

SUMMARY:
The purpose of this study is to evaluate the visual quality and function of pseudophakic patients.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Pseudophakic patients who have been bilaterally implanted with the same type of intraocular lenses in both eyes
* Ability to understand, read and write English to give consent and complete the study questionnaires
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures and study visits
* Signed informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization
* Other protocol-defined inclusion criteria might apply

Exclusion Criteria:

* Any ocular pathology of clinical significance, as determined by the investigator, that may affect visual outcomes or influence subjective ocular/visual symptoms
* Patient is pregnant or is lactating
* Concurrent participation or participation within 30 days prior in any other clinical trial
* Other protocol-defined exclusion criteria might apply

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bilaterally-implanted pseudophakic subjects over 22 years of age who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Daniel Chang, M.D., Bakersfield, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pseudophakic: .
  Administration of patient self assessment
Period: Overall Study
Arm/Group | Pseudophakic
Started | 301
Completed | 296
Not Completed | 5
Not completed — Failed to meet inclusion criteria | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pseudophakic
Number analyzed (Participants) | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.79 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 102

OUTCOME MEASURES:

1. Primary Outcome: Use of Corrective Visual Aids (i.e., Spectacles, Contact Lenses) Post Intraocular Lens (IOL) Surgery
Description: Patients will be assessed at a baseline visit and a visit 1 week later to determine their use of corrective visual aids (i.e., spectacles, contact lenses) post Intraocular Lens (IOL) surgery.
Time Frame: Baseline and 1 week
Population: Of the 295 participants who provided data for this analysis (monofocal participants , n=138; accommodating participants, n=34; and multifocal participants, n=123), corrective visual aids (i.e., spectacles, contact lenses) post intraocular lens (IOL) surgery were required by 88 participants.
Measure: Number; unit: participants
Arm/Group | Pseudophakic
Number analyzed (Participants) | 295
participants
  Monofocal participants requiring visual aids | 71
  Accommodating participants requiring visual aids | 8
  Multifocal participants requiring visual aids | 9

ADVERSE EVENTS:
Arm/Group | Pseudophakic
Serious Adverse Events (participants affected / at risk) | 0/296
Other Adverse Events (participants affected / at risk) | 0/296

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other